CLINICAL TRIAL: NCT02690350
Title: A Phase 1, Open-label, Two-part, Safety and Tolerability Study of U3-1784 in Patients With Advanced Solid Tumours
Brief Title: An Open Study Assessing the Safety and Tolerability of U3-1784
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Program discontinued for business reasons (not safety).
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: U31784-A-E101; 2015-002670-20 (EudraCT Number)
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Advanced Solid Tumors; Hepatocellular Cancer (HCC)
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, three cohorts
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 U3-1784 2.5 mg/kg (Experimental): U3-1784 (2.5 mg/kg) by intravenous infusion, along with colestyramine or equivalent if clinically indicated
  Interventions: Drug: U3-1784
- Cohort 2 U3-1784 3.75 mg/kg (Experimental): U3-1784 (3.75 mg/kg) by intravenous infusion, along with colestyramine or equivalent if clinically indicated
  Interventions: Drug: U3-1784
- Cohort 3 U3-1784 5.6 mg/kg (Experimental): U3-1784 (5.6 mg/kg) by intravenous infusion, along with colestyramine or equivalent if clinically indicated
  Interventions: Drug: U3-1784

INTERVENTIONS:
Drug: U3-1784 — Solution for solution in 5% dextrose for infusion, intravenously administered every 2 weeks (q2w) as a 250 mL IV, along with colestyramine or equivalent if clinically indicated
  Other Names: Experimental product

SUMMARY:
The main objectives of the trial are:

* To evaluate the safety and tolerability of U3-1784 in patients with advanced solid tumours
* To determine the maximum tolerated dose (MTD) and or establish the safety and tolerability of the maximum administered dose (MAD) of U3-1784

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Patients with histologically or cytologically confirmed advanced solid tumours refractory to, intolerant of, or not eligible for standard treatment, or who decline standard therapy, or for whom no therapy with curative intent is available
* Part 2: Patients with histologically or cytologically confirmed HCC refractory to, intolerant of, or not eligible for standard treatment, or who decline standard therapy, or for whom no therapy with curative intent is available. If emerging Part 1 data suggest that a particular tumour type or specific tumour histology might be responsive to treatment, then patients with this tumour type or histology will also be included in Part 2 of the study.
* Male or female patients, 18 years of age or older.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment.
* Males and females of childbearing potential are permitted in the study so long as they consent to avoid getting their partner pregnant or becoming pregnant, respectively, by using a highly effective contraception method, as described below, throughout the study and for up to 90 days after completion. Highly effective methods of contraception include: hormonal methods associated with inhibition of ovulation, intrauterine device; surgical sterilization (including partner's vasectomy) or sexual abstinence, if this is the preferred and usual lifestyle of the subject. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year Eastern Cooperative Oncology Group performance status ≤ 1.
* Life expectancy of greater than 3 months.
* Ability to understand and the willingness to sign a written informed consent form.
* Measurable or evaluable disease as defined by RECIST Version 1.1 in Part 1 of the study (patients included in Part 2 will be required to have measurable disease). The measurable lesion in HCC patients should not be one that has been previously treated by loco-regional therapies (e.g. TACE, RFA) unless this lesion has progressed and there is evidence of new, measurable, enhancement on dynamic imaging.
* Patient has 1 of the following available for pharmacodynamic analyses:
* Archived diagnostic or freshly obtained formalin-fixed paraffin embedded or frozen tumour tissue
* Tumour tissue biopsy collected prior to study drug administration
* Patient has adequate bone marrow, renal, and hepatic function as follows:
* Haemoglobin: ≥ 90 g/L
* Absolute Neutrophil Count: ≥ 1.5 × 109/L
* Platelets: ≥ 100 × 109/L (Part 1); ≥ 75 × 109/L (Part 2)
* Total Bilirubin: ≤ 1.5 × upper limit of normal (ULN)
* AST (SGOT)/ALT (SGPT): ≤ 2.5 × institutional ULN
* Prothrombin Time (PT)/International Normalised Ratio (INR): ≤ 1.5 (patients on anticoagulants will have PT and INR as determined by the Investigator)
* Serum creatinine: ≤ 1.5 × ULN or Creatinine Clearance (calculated from serum creatinine using Cockcroft-Gault formula) ≥ 60 mL/min for patients with creatinine levels above institutional normal

Exclusion Criteria:

* Patient has received anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational therapy or loco-regional therapy within a period of 21 days prior to Study Day 1 (6 weeks for nitrosureas or mitomycin C). Prior and concurrent use of hormone replacement therapy, use of gonadotropin-releasing hormone modulators for prostate cancer, and use of somatostatin analogues for neuroendocrine tumours are permitted.
* Patient has unresolved clinically significant toxicities from prior anticancer therapy, defined as any National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03; Grade 2 or higher, apart from alopecia.
* Patients with heart failure (New York Heart Association > Class II) within 6 months prior to study entry; symptomatic coronary artery disease; clinically significant cardiac arrhythmia defined as ≥ Grade 3 to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03; uncontrolled hypertension, myocardial infarction occurring within 6 months prior to study entry.
* Patient has active clinically serious infection defined as ≥ Grade 3 to NCI CTCAE, Version 4.03.
* Patients with clinically significant pericardial effusions, pleural effusions or ascites.
* Patient has had another active malignancy within the past 3 years except for nonmelanoma carcinoma of the skin, cervical carcinoma in situ, and superficial bladder tumours.
* Patient has had major surgery within 4 weeks before enrolment.
* Patient has known hypersensitivity to colestyramine (or any of its excipients) or history of hypersensitivity/allergic reactions attributed to other monoclonal antibodies
* Patients with complete biliary obstruction
* Lactating women

Additional exclusion criteria for HCC patients included in Part 1 and Part 2:

* Concomitant interferon therapy or therapies for active Hepatitis C Virus infection.
* Patient has history of liver transplant.
* Patient has Child-Pugh B-C cirrhotic status based on clinical findings and laboratory results during screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events | within 1 year
  Treatment emergent adverse events (TEAEs) are systematically collected - clinically significant changes in laboratory values are recorded as TEAEs in system organ class: Investigations
Number of Patients with Dose-Limiting Toxicities (DLTs) | from start of treatment until trial termination (within 2 months)

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) | within 2 months
Time to Cmax (Tmax) | within 2 months
Area Under the Curve to the Last Quantifiable Measure (AUClast)[ | within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Martinez, PhD, Study Director — Daiichi Sankyo UK Ltd.
Locations (4):
- United Kingdom (4):
  - Glasgow, Lanarkshire
  - The Royal Marsden Hospital, Sutton, Surrey
  - Guy's Hospital, London
  - The Christie NHS Foundation Trust, Manchester